CLINICAL TRIAL: NCT01328379
Title: Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Safety and Efficacy of Two Doses of Oral Dalfampridine Extended Release Tablets (5 mg and 10 mg Twice Daily) in Patients With Multiple Sclerosis
Brief Title: Study of Fampridine-ER Tablets in Patients With Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DER-401
Record Dates: First submitted 2011-03-29; First posted 2011-04-04 (Estimated); Results first posted 2013-08-13 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dalfampridine-ER 5mg (Active Comparator): 5mg, twice daily
  Interventions: Drug: Dalfampridine-ER 5mg
- Dalfampridine-ER 10mg (Active Comparator): 10mg, twice daily
  Interventions: Drug: Dalfampridine-ER 10mg
- Placebo (Placebo Comparator): placebo, twice daily
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dalfampridine-ER 5mg — 5mg, twice daily
  Other Names: Fampridine, Dalfampridine, Ampyra
  Arms: Dalfampridine-ER 5mg
Drug: Dalfampridine-ER 10mg — 10mg, twice daily
  Other Names: Fampridine, Dalfampridine, Ampyra
  Arms: Dalfampridine-ER 10mg
Other: Placebo — placebo, twice daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of a lower dose of dalfampridine extended release tablets compared to the currently approved dose in improving walking in Multiple Sclerosis (MS) patients.

DETAILED DESCRIPTION:
The current study is designed as a prospective placebo-controlled trial to investigate the safety and efficacy of a lower dose of dalfampridine extended release tablets (5 mg twice daily) compared to the approved commercial dose of 10 mg twice daily in improving walking in MS patients during a four-week period of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient has clinically definite Multiple Sclerosis as defined by the MacDonald Criteria.
* Patient must be 18 to 70 years of age, inclusive (i.e. on or after their 18th birthday, up to the day before their 71st birthday at the Screening Visit).
* Patient who has previously taken Ampyra® or dalfampridine (fampridine or 4 aminopyridine; 4-AP) in any formulation (including compounded), must have withdrawn from the drug for at least one month prior to the Screening Visit.
* Patient must be mentally competent to understand and sign the Internal Review Board (IRB)-approved informed consent prior to the performance of any study-specific procedures.
* Patient is able to perform all the required study procedures.
* In the judgement of the Investigator, the patient has MS-related walking impairment but has sufficient ambulatory ability to be able to complete two trials of the Timed 25 Foot Walk (T25FW) at the screening Visit and every study visit thereafter, with the two trials completed within 5 minutes of one another and in accordance with the specific instructions provided by the National Multiple Sclerosis Society MS Functional Composite Manual.
* Patient who is female and of childbearing potential (see Exclusion Criterion 1 for definition) must have a negative urine pregnancy test at the Screening Visit.

Exclusion Criteria:

* Patient is a female of childbearing potential (i.e., has not had a hysterectomy or bilateral oophorectomy, or is not at least two years postmenopausal), engaged in active heterosexual relations and is not using one of the following birth control methods: tubal ligation, implantable contraception device, oral, patch or injectable contraceptive, double barrier method, or sexual activity restricted to vasectomized partner.
* Patient is pregnant or breastfeeding.
* Patient has any history of seizures.
* Patient has moderate or severe renal impairment as defined by a calculated creatinine clearance of ≤ 50 mL/minute.
* Patient has active urinary tract infection (UTI) at Screening or within the 4 weeks before Screening.
* Patient has had an onset (as assessed by the treating physician) of an MS exacerbation within 60 days prior to the Screening Visit.
* Patient has started on a concomitant prescription medication regimen within the last three weeks, and/or their concomitant medication regimen is expected to change during the course of the study.
* Patient has received cyclophosphamide (Cytoxan) or mitoxantrone (Novantrone) for MS treatment within six months prior to the Screening Visit.
* Patient has started a treatment regimen of Betaseron, Avonex, Copaxone, Rebif, Tysabri, Extavia or Gilenya™ within 90 days prior to the Screening Visit or has had any change in the dosing regimen of these drugs within 30 days prior to the Screening Visit.
* Patient has received corticosteroids (other than topical preparations) within 30 days prior to the Screening Visit and/or is expected to receive regularly scheduled corticosteroid treatment during the course of the study.
* Patient has been administered botulinum toxin in the lower extremities within six months prior to the Screening Visit and/or is expected to receive botulinum toxin in the lower extremities during the course of the study.
* Patient has a known allergy to pyridine-containing substances or any of the inactive ingredients of the dalfampridine tablet (colloidal silicon dioxide, hydroxypropyl methylcellulose, magnesium stearate, microcrystalline cellulose, polyethylene glycol, and titanium dioxide).
* Patient has a history of drug or alcohol abuse within the past year.
* Patient has clinically significant abnormal laboratory values.
* Patient has angina, uncontrolled hypertension, clinically significant cardiac arrhythmias, or any other clinically significant cardiovascular abnormality.
* Patient has any medical condition (including psychiatric disease)that would interfere with the interpretation of the study results or the conduct of the study.
* Patient has participated in an investigational trial 30 days prior to Screening Visit or plans to enroll in another investigational trial at any time during this study. Non-drug (i.e. observational, registry) and non- medical device trials are allowed.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2011-03; Primary Completion 2012-04 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew R. Blight, PhD, Study Director — Acorda Therapeutics; Mark Agius, MD, Principal Investigator — University of California, Davis; Angela Applebee, MD, Principal Investigator — University of Vermont Medical Center; S. A Azizi, MD, PhD, Principal Investigator — Temple University Hospital; Francois Bethoux, MD, Principal Investigator — The Cleveland Clinic; Christopher Bever, Jr., MD, Principal Investigator — University of Maryland, Maryland Center for Multiple Sclerosis; Eric Borresen, MD, Principal Investigator — Metrolina Medical Research; Aaron Boster, MD, Principal Investigator — Ohio State University, Columbus; Ann Camac, MD, Principal Investigator — Lahey Clinic; Mark Cascione, MD, Principal Investigator — Axiom Clinical Research of Florida; Jane Chan, MD, Principal Investigator — US Department of Veterans Affairs; Warren Chumley, MD, Principal Investigator — Associates in Neurology, PSC; Joanna Cooper, MD, Principal Investigator — Alta Bates Summit Medical Center; Joy Derwenskus, DO, Principal Investigator — Northwestern University; Adam DiDio, MD, Principal Investigator — Suncoast Neuroscience Associates, Inc.; Dennis Dietrich, MD, Principal Investigator — Advanced Neurology Specialists; Geoffery Eubank, MD, Principal Investigator — Neurological Research Institute; Steven Freedman, MD, Principal Investigator — Raleigh Neurology Associates; Daniel Giang, MD, Principal Investigator — Loma Linda University Medical Center; Lawrence Goldstick, MD, Principal Investigator — Neurology Specialists, Inc.; Andrew Goodman, MD, Principal Investigator — University of Rochester; Mark Gudesblatt, MD, Principal Investigator — Comprehensive Multiple Sclerosis Care Center at South Shore Neurologic Associates, P.C.; Barry Hendin, MD, Principal Investigator — Phoenix Neurological Associates, LTD; Craig Herrman, MD, Principal Investigator — Josephson Wallack Munshower Neurology, PC; William Honeycutt, MD, Principal Investigator — Neurology Associates, PA; Bruce Hughes, MD, Principal Investigator — Ruan Neurology Clinical Research Center; Samuel Hunter, MD, PhD, Principal Investigator — Advanced Neurosciences Institute; George Hutton, MD, Principal Investigator — Maxine Mesinger Multiple Sclerosis Clinic; Baylor College of Medicine; Dina Jacobs, MD, Principal Investigator — University of Pennsylvania; Todd Janus, MD, PhD, Principal Investigator — Iowa Health Des Moines; Omar Khan, MD, Principal Investigator — Wayne State University; Bhupendra Khatri, MD, Principal Investigator — Aurora Saint Luke's Medical Center; Kiren Kresa-Reahl, MD, Principal Investigator — Charleston Area Medical Center Health Education and Research Institute, Inc.; Christopher LaGanke, MD, Principal Investigator — North Central Neurology Associates, PC; Sharon Lynch, MD, Principal Investigator — University of Kansas Medical Center; Michele Mass, MD, Principal Investigator — Oregon Health and Science University; David Mattson, MD, PhD, Principal Investigator — Indiana University; Angeli Mayadev, MD, Principal Investigator — Swedish Neuroscience Institute; Donald Negroski, MD, Principal Investigator — Negroski, Stein, Sutherland and Hanes Neurology; Stephen Newman, MD, Principal Investigator — Island Neurological Associates, PC; Gabriel Pardo, MD, Principal Investigator — Mercy Multiple Sclerosis Center of Oklahoma Mercy Neuroscience Institute; C. Fish Greenfield, MD, Principal Investigator — Texas Neurology, PA; Rekha Pillai, MD, Principal Investigator — Neurology Clinic, PC; T. Hemanth Rao, MD, Principal Investigator — The Neurological Institute, PA; Syed Rizvi, MD, Principal Investigator — Rhode Island Hospital; Matthew Roller, MD, Principal Investigator — Altru Health System Research Center; Michael Rossen, MD, PhD, Principal Investigator — Springfield Neurology Associates, LLC; Alan Schulman, MD, Principal Investigator — Neurological Associates; James S Shafer, MD, Principal Investigator — The Multiple Sclerosis Center of Vero Beach; Jatin Shah, MD, Principal Investigator — Arizona Neurological Institute; William Sheremata, MD, Principal Investigator — University of Miami School of Medicine, Dept. of Neurology; Brian Steingo, MD, Principal Investigator — Neurological Associates; James Storey, Jr, MD, Principal Investigator — Upstate Clinical Research, LLC; Ben Thrower, MD, Principal Investigator — Shepherd Center, Inc.; Carlo Tornatore, MD, Principal Investigator — Georgetown University Hospital; K A Lloyd, MD, Principal Investigator — Hampton Roads Neurology; Anthony Turel, Jr, MD, Principal Investigator — The Pennsylvania State University, Milton S. Hershey Medical Center; Sibyl E Wray, MD, Principal Investigator — Sibyl E. Wray, MD, Neurology, PC; Daniel Wynn, MD, Principal Investigator — Consultants in Neurology Ltd.; Robert Yapundich, MD, Principal Investigator — Unifour Medical Research, LLC
Locations (70):
- United States (70):
  - North Central Neurology Associates, PC, Cullman, Alabama
  - Phoenix Neurological Associates, Ltd, Phoenix, Arizona
  - Arizona Neurological Institute, Sun City, Arizona
  - Clinical Research Advantage Inc., Tempe, Arizona
  - Sutter East Bay Physicians Medical Foundation, Berkeley, California
  - Neuro-Pain Medical Center, Inc., Fresno, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Collaborative NeuroScience Network, Inc., Long Beach, California
  - University of California Davis Medical Center, Sacramento, California
  - Mount Sinai Rehabilitation Hospital, Hartford, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Neurology Associates, PA, Maitland, Florida
  - University of Miami School of Medicine, Dept. of Neurology, Miami, Florida
  - Neurological Associates, Pompano Beach, Florida
  - Neurologique Foundation, Inc., Ponte Vedra, Florida
  - Negroski, Sutherland and Hanes Neurology, Sarasota, Florida
  - Suncoast Neuroscience Associates, Inc., St. Petersburg, Florida
  - Tallahassee Neurological Clinic, PA, Tallahassee, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - The Multiple Sclerosis Center of Vero Beach, Vero Beach, Florida
  - Sheperd Center, Inc., Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Consultants in Neurology Ltd., Northbrook, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Josephson Wallack Munshower Neurology, PC, Indianapolis, Indiana
  - Methodist Plaza Specialty, Des Moines, Iowa
  - Ruan Neurology Clinic and Research Center, Des Moines, Iowa
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Associates in Neurology, PSC, Lexington, Kentucky
  - University of Maryland, Maryland Center for Multiple Sclerosis, Baltimore, Maryland
  - Lahey Clinic, Lexington, Massachusetts
  - Springfield Neurology Associates, LLC, Springfield, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Advanced Neurology Specialists, Great Falls, Montana
  - Veterans Administration Sierra Neveda Health Care System, Reno, Nevada
  - Upstate Clinical Research, LLC, Albany, New York
  - NYU Langone Medical Center MS Comprehensive Care Center, New York, New York
  - Comprehensive Multiple Sclerosis Care Center at South Shore Neurologic Associates, Patchogue, New York
  - Island Neurological Associates, PC, Plainview, New York
  - University of Rochester Medical Center, Rochester, New York
  - PMG Research of Charlotte, Charlotte, North Carolina
  - The Neurological Institute, PA, Charlotte, North Carolina
  - PMG Research of Hickory, LLC, Hickory, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Altru Health System Clinic, Grand Forks, North Dakota
  - Northern Ohio Neuroscience, LLC, Bellevue, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Neurological Research Institute, Columbus, Ohio
  - Ohio State University, Columbus, Columbus, Ohio
  - Neurology Specialists, Inc., Dayton, Ohio
  - OMRF Multiple Sclerosis Center of Excellence, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Providence Multiple Sclerosis Center, Portland, Oregon
  - The Pennsylvania State University, Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - The Neurology Foundation, Inc., Providence, Rhode Island
  - Wesley Neurology Clinic, PC, Cordova, Tennessee
  - Advanced Neurosciences Institute, Franklin, Tennessee
  - Sibyl E. Wray, MD, Neurology, PC, Knoxville, Tennessee
  - Texas Neurology, PA, Dallas, Texas
  - Kelsey-Seybold Clinic, Houston, Texas
  - Maxine Mesinger Multiple Sclerosis Clinic; Baylor College of Medicine, Houston, Texas
  - Fletcher Allen Health Care, Burlington, Vermont
  - Hampton Roads Neurology, Newport News, Virginia
  - Neurological Associates, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Swedish Neuroscience Institute, Seattle, Washington
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Applebee A, Goodman AD, Mayadev AS, Bethoux F, Goldman MD, Klingler M, Blight AR, Carrazana EJ. Effects of Dalfampridine Extended-release Tablets on 6-minute Walk Distance in Patients With Multiple Sclerosis: A Post Hoc Analysis of a Double-blind, Placebo-controlled Trial. Clin Ther. 2015 Dec 1;37(12):2780-7. doi: 10.1016/j.clinthera.2015.10.014. Epub 2015 Nov 10. PMID 26565077
- [Derived] Kantor D, Chancellor MB, Snell CW, Henney HR 3rd, Rabinowicz AL. Assessment of confirmed urinary tract infection in patients treated with dalfampridine for multiple sclerosis. Postgrad Med. 2015 Mar;127(2):218-22. doi: 10.1080/00325481.2015.1000229. Epub 2015 Jan 6. PMID 25560174

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were to be enrolled at a minimum of 60 investigational centers in the United States until a minimum of 405 patients had been randomized.
Period: Overall Study
Arm/Group | Placebo | Dalfampridine-ER 5mg | Dalfampridine-ER 10mg
Started | 143 | 144 | 143
Completed | 142 | 144 | 143
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: All randomized patients who took at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dalfampridine-ER 5mg | Dalfampridine-ER 10mg | Total
Number analyzed (Participants) | 142 | 144 | 143 | 429
Age Continuous [Mean (Standard Deviation); unit: years] | 52.2 (0.83) | 52.2 (0.77) | 53.4 (0.79) | 52.6 (0.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 102 | 98 | 300
  Male | 42 | 42 | 45 | 129
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 7 | 3 | 20
  Not Hispanic or Latino | 132 | 137 | 140 | 409
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Walking Speed Near Maximum Plasma Concentration at Steady State (CmaxSS) of Placebo and Dalfampridine-ER (5mg and 10mg), Using the Timed 25 Foot Walk (T25FW).
Description: The T25FW test is a quantitative measure of ambulatory function that is widely used by MS specialists to assess the global impact of the disease and its progression on the patient's physical disability.
  A patient will stand with the toes of his/her shoes on the starting line (identified by a taped mark on the floor) and timing will begin when any part of the patient's foot crosses the tape. Timing will end when any part of the patient's foot crosses the finish line (identified by a taped mark on the floor). Time will be recorded in seconds and rounded to the nearest tenth of a second using a stopwatch provided for this study.
Time Frame: Baseline Visit 1 (double-blind study day 1) and approximately 3-4 hours post dose at Visit 3 (end of double-blind week 4)
Population: Full Analysis Population (FAP): All randomized patients who took at least one dose of double-blind investigational medication and who have a baseline Timed 25 Foot Walk (T25FW) assessment and at least one post-baseline T25FW assessment.
Measure: Mean (Standard Error); unit: feet per second
Arm/Group | Placebo | Dalfampridine-ER 5mg | Dalfampridine-ER 10mg
Number analyzed (Participants) | 136 | 143 | 136
feet per second | 0.363 (0.0511) | 0.423 (0.0470) | 0.478 (0.0569)
Statistical Analysis 1: Comparison: Placebo vs Dalfampridine-ER 5mg; dalfampridine-ER 5mg twice daily vs. placebo twice daily: Change from baseline in walking speed at Approximately CmaxSS at Visit 3; Test type: Superiority or Other; p = 0.457, ANOVA — To demonstrate study sensitivity with respect to efficacy and maintain an overall alpha level ≤ 0.05, a stepwise procedure was performed; ANOVA Model: Change from Baseline in Walking Speed - dependent variable and Baseline Walking Speed and Treatment - independent variables; least squares mean = 0.054, 95% CI 2-sided [-0.088 to 0.196], Standard Error of Mean 0.0724
Statistical Analysis 2: Comparison: Placebo vs Dalfampridine-ER 10mg; dalfampridine-ER 10mg twice daily vs. placebo twice daily: Change from baseline in walking speed at Approximately CmaxSS at Visit 3; Test type: Superiority or Other; p = 0.107, ANOVA; [statistical method as in outcome 1, analysis 1]; least squares mean = 0.118, 95% CI 2-sided [-0.026 to 0.262], Standard Error of Mean 0.0732
Statistical Analysis 3: Comparison: Dalfampridine-ER 5mg vs Dalfampridine-ER 10mg; dalfampridine-ER 5mg twice daily vs. dalfampridine-ER 10mg twice daily: Change from baseline in walking speed at Approximately CmaxSS at Visit 3; Test type: Superiority or Other; p = 0.375, ANOVA; [statistical method as in outcome 1, analysis 1]; least squares mean = 0.064, 95% CI 2-sided [-0.078 to 0.207], Standard Error of Mean 0.0724

2. Secondary Outcome: Change From Baseline in Walking Speed Near Minimum Plasma Concentration at Steady State (CminSS) of Placebo, Dalfampridine-ER (5mg and 10mg), Using the Timed 25 Foot Walk (T25FW).
Description: as for outcome 1
Time Frame: Baseline Visit 1 (double-blind study day 1) and approximately 12 hours post dose at Visit 3 (end of double-blind week 4)
Population: Full Analysis Population
Measure: Mean (Standard Error); unit: feet per second
Arm/Group | Placebo | Dalfampridine-ER 5mg | Dalfampridine-ER 10mg
Number analyzed (Participants) | 136 | 143 | 136
feet per second | 0.301 (0.0496) | 0.296 (0.0429) | 0.391 (0.0513)
Statistical Analysis 1: Comparison: Placebo vs Dalfampridine-ER 5mg; dalfampridine-ER 5mg twice daily vs. placebo twice daily: Change from baseline in walking speed at Approximately CminSS at Visit 3; Test type: Superiority or Other; p = 0.832, ANOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Least Squares Mean = -0.014, 95% CI 2-sided [-0.145 to 0.117], Standard Error of Mean 0.0666
Statistical Analysis 2: Comparison: Placebo vs Dalfampridine-ER 10mg; dalfampridine-ER 10mg twice daily vs. placebo twice daily: Change from baseline in walking speed at Approximately CminSS at Visit 3; Test type: Superiority or Other; p = 0.167, ANOVA; [statistical method as in outcome 1, analysis 1]; Least Squares Mean = 0.093, 95% CI 2-sided [-0.039 to 0.226], Standard Error of Mean 0.0674
Statistical Analysis 3: Comparison: Dalfampridine-ER 5mg vs Dalfampridine-ER 10mg; dalfampridine-ER 5mg twice daily vs. dalfampridine-ER 10mg twice daily: Change from baseline in walking speed at Approximately CminSS at Visit 3; Test type: Superiority or Other; p = 0.108, ANOVA; [statistical method as in outcome 1, analysis 1]; Least Squares Mean = 0.107, 95% CI 2-sided [-0.024 to 0.238], Standard Error of Mean 0.0666

3. Secondary Outcome: Change From Baseline in 12-item MS Walking Scale (MSWS-12) at Visit 3
Description: The MSWS-12 is a multi-item rating scale that asks patients to rate limitations of their mobility due to MS during the preceding two weeks on a 5-point scale (from 1= not at all to 5=extremely). The scale assesses a range of activities of daily life that rely on walking, such as climbing stairs, moving around the home and walking distances outdoors. The MSWS-12 also addresses the quality of walking, with questions on the smoothness, speed, distance, effort, and mental concentration involved in walking, as well as the need for assistive devices.
  For each visit, the MSWS-12 score was calculated by summing the 12 components and transforming into a scale with a range of 0 to 100.
  MSWS-12 Score = 100 * [(Sum of Items 1-12) - 12]/48
Time Frame: Baseline Visit 1 (double-blind study day 1) and Visit 3 (end of double-blind week 4)
Population: Full Analysis Population
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Dalfampridine-ER 5mg | Dalfampridine-ER 10mg
Number analyzed (Participants) | 136 | 143 | 136
scores on a scale | -8.35 (1.774) | -9.73 (1.741) | -11.10 (1.818)
Statistical Analysis 1: Comparison: Placebo vs Dalfampridine-ER 5mg; dalfampridine-ER 5mg twice daily vs. placebo twice daily: Change from baseline in MSWS-12 at visit 3; Test type: Superiority or Other; p = 0.866, ANOVA; ANOVA model with change from baseline in MSWS-12 Score as the dependent variable and baseline MSWS-12 Score and treatment as the independent variables; Lease Squares Mean = -0.40, 95% CI 2-sided [-5.05 to 4.25], Standard Error of Mean 2.367
Statistical Analysis 2: Comparison: Placebo vs Dalfampridine-ER 10mg; dalfampridine-ER 10mg twice daily vs. placebo twice daily: Change from baseline in MSWS-12 at visit 3; Test type: Superiority or Other; p = 0.286, ANOVA; [statistical method as in outcome 3, analysis 1]; Least Squares Mean = -2.56, 95% CI 2-sided [-7.26 to 2.15], Standard Error of Mean 2.393
Statistical Analysis 3: Comparison: Dalfampridine-ER 5mg vs Dalfampridine-ER 10mg; dalfampridine-ER 5mg twice daily vs. dalfampridine-ER 10mg twice daily: Change from baseline in MSWS-12 at visit 3; Test type: Superiority or Other; p = 0.362, ANOVA; [statistical method as in outcome 3, analysis 1]; Least Squares Mean = -2.16, 95% CI 2-sided [-6.81 to 2.49], Standard Error of Mean 2.366

4. Secondary Outcome: Change From Baseline in MSWS-12 at Visit 2
Description: as for outcome 3
Time Frame: Visit 1 (Baseline) and Visit 2 (start of third week double-blind treatment period )
Population: Full Analysis Population
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Dalfampridine-ER 5mg | Dalfampridine-ER 10mg
Number analyzed (Participants) | 136 | 142 | 136
scores on a scale | -9.48 (1.713) | -9.54 (1.526) | -10.04 (1.817)
Statistical Analysis 1: Comparison: Placebo vs Dalfampridine-ER 5mg; dalfampridine-ER 5mg twice daily vs. placebo twice daily: Change from baseline in MSWS-12 at visit 2; Test type: Superiority or Other; p = 0.708, ANOVA; [statistical method as in outcome 3, analysis 1]; Least Squares Mean = 0.84, 95% CI 2-sided [-3.56 to 5.24], Standard Error of Mean 2.237
Statistical Analysis 2: Comparison: Placebo vs Dalfampridine-ER 10mg; dalfampridine-ER 10mg twice daily vs. placebo twice daily: Change from baseline in MSWS-12 at visit 2; Test type: Superiority or Other; p = 0.868, ANOVA; [statistical method as in outcome 3, analysis 1]; Least Squares Mean = -0.38, 95% CI 2-sided [-4.81 to 4.06], Standard Error of Mean 2.258
Statistical Analysis 3: Comparison: Dalfampridine-ER 5mg vs Dalfampridine-ER 10mg; dalfampridine-ER 5mg twice daily vs. dalfampridine-ER 10mg twice daily: Change from baseline in MSWS-12 at visit 2; Test type: Superiority or Other; p = 0.588, ANOVA; [statistical method as in outcome 3, analysis 1]; Least Squares Mean = -1.21, 95% CI 2-sided [-5.61 to 3.18], Standard Error of Mean 2.236

5. Secondary Outcome: Change From Baseline in Six-Minute Walk Distance at Visit 2
Description: The Six-Minute Walk, a test of endurance, measures the distance that a patient can walk in a period of 6 minutes. Six-minute walk distance will be reported in feet.
Time Frame: Visit 1 (Baseline) and Visit 2 (start of third week double-blind treatment period )
Population: Full Analysis Population
Measure: Mean (Standard Error); unit: Feet
Arm/Group | Placebo | Dalfampridine-ER 5mg | Dalfampridine-ER 10mg
Number analyzed (Participants) | 49 | 53 | 51
Feet | 41.7 (23.36) | 76.8 (27.31) | 128.6 (21.66)
Statistical Analysis 1: Comparison: Placebo vs Dalfampridine-ER 5mg; dalfampridine-ER 5mg twice daily vs. placebo twice daily: Change from baseline in Six-Minute Walk Distance at visit 2; Test type: Superiority or Other; p = 0.308, ANOVA; Change from Baseline in Six-Minute Walk Distance as dependent variable and Baseline Six-Minute Walk Distance and Treatment as independent variables; Least Squares Mean = 35.4, 95% CI 2-sided [-33.0 to 103.7], Standard Error of Mean 34.57
Statistical Analysis 2: Comparison: Placebo vs Dalfampridine-ER 10mg; dalfampridine-ER 10mg twice daily vs. placebo twice daily: Change from baseline in Six-Minute Walk Distance at visit 2; Test type: Superiority or Other; p = 0.014, ANOVA; [statistical method as in outcome 5, analysis 1]; Least Squares Mean = 87.1, 95% CI 2-sided [18.2 to 156.1], Standard Error of Mean 34.90
Statistical Analysis 3: Comparison: Dalfampridine-ER 5mg vs Dalfampridine-ER 10mg; dalfampridine-ER 5mg twice daily vs. dalfampridine-ER 10mg twice daily: Change from baseline in Six-Minute Walk Distance at visit 2; Test type: Superiority or Other; p = 0.133, ANOVA; [statistical method as in outcome 5, analysis 1]; Least Squares Mean = 51.7, 95% CI 2-sided [-15.9 to 119.3], Standard Error of Mean 34.21

6. Secondary Outcome: Change From Baseline in EuroQol Group 5 Dimensions (EQ-5D) Scores at Visit 3.
Description: Patients completed a brief, generic health status questionnaire: The five specific dimensional scores value patients' health related to mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. Each question has 3 distinguishable choices that can be analyzed using a 3-point scale (i.e. 1 = no problem, 2=some problems and 3= extreme problems).
  A response of 1 indicates that the patient has no problem with the dimension tested and a response of 3 indicates that the patient has extreme problems with the dimension tested. For each visit, the average score of 5 dimensions was calculated by averaging the scores of 5 dimensions. EQ-5D final score ranges from 1-3.
Time Frame: Baseline Visit 1 (double-blind study day 1) and Visit 3 (end of double-blind week 4)
Population: Full Analysis Population
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Dalfampridine-ER 5mg | Dalfampridine-ER 10mg
Number analyzed (Participants) | 132 | 139 | 126
units on a scale | -0.07 (0.023) | -0.05 (0.020) | -0.07 (0.024)
Statistical Analysis 1: Comparison: Placebo vs Dalfampridine-ER 5mg; dalfampridine-ER 5mg twice daily vs. placebo twice daily: Change from baseline in Average EQ-5D score at Visit 3; Test type: Superiority or Other; p = 0.320, ANOVA; ANOVA model with change from baseline score as the dependant variable and baseline score and treatment as the independent variables; Least Squares Mean = 0.0, 95% CI 2-sided [-0.0 to 0.1], Standard Error of Mean 0.03
Statistical Analysis 2: Comparison: Placebo vs Dalfampridine-ER 10mg; dalfampridine-ER 10mg twice daily vs. placebo twice daily: Change from baseline in Average EQ-5D score at Visit 3; Test type: Superiority or Other; p = 0.734, ANOVA; [statistical method as in outcome 6, analysis 1]; Least Squares Mean = -0.0, 95% CI 2-sided [-0.1 to 0.0], Standard Error of Mean 0.03
Statistical Analysis 3: Comparison: Dalfampridine-ER 5mg vs Dalfampridine-ER 10mg; dalfampridine-ER 5mg twice daily vs. dalfampridine-ER 10mg twice daily: Change from baseline in Average EQ-5D score at Visit 3; Test type: Superiority or Other; p = 0.185, ANOVA; [statistical method as in outcome 6, analysis 1]; Least Squares Mean = -0.0, 95% CI 2-sided [-0.1 to 0.0], Standard Error of Mean 0.03

7. Secondary Outcome: Change From Baseline in EQ-5D Visual Analogue Self-rating (VAS) Score at Visit 3.
Description: The EQ-5D is a brief questionnaire that asks patients to rate general state of health. The VAS score rates the general state of health of a patient with 100 for the best imaginable health state and 0 for the worst imaginable health state.
Time Frame: Baseline Visit 1 (double-blind study day 1) and Visit 3 (end of double-blind week 4)
Population: Full Analysis Population. The number of participants analyzed corresponds with number of subjects who completed the questionnaire in each treatment group.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Dalfampridine-ER 5mg | Dalfampridine-ER 10mg
Number analyzed (Participants) | 131 | 139 | 127
units on a scale | 7.0 (1.43) | 2.6 (1.53) | 4.2 (1.48)
Statistical Analysis 1: Comparison: Placebo vs Dalfampridine-ER 5mg; dalfampridine-ER 5mg twice daily vs. placebo twice daily: Change from baseline in EQ-5D VAS score at Visit 3; Test type: Superiority or Other; p = 0.055, ANOVA; [statistical method as in outcome 6, analysis 1]; Least Squares Mean = -3.4, 95% CI 2-sided [-7.0 to 0.1], Standard Error of Mean 1.79
Statistical Analysis 2: Comparison: Placebo vs Dalfampridine-ER 10mg; dalfampridine-ER 10mg twice daily vs. placebo twice daily: Change from baseline in EQ-5D VAS score at Visit 3; Test type: Superiority or Other; p = 0.530, ANOVA; [statistical method as in outcome 6, analysis 1]; Least Squares Mean = -1.2, 95% CI 2-sided [-4.7 to 2.4], Standard Error of Mean 1.83
Statistical Analysis 3: Comparison: Dalfampridine-ER 5mg vs Dalfampridine-ER 10mg; dalfampridine-ER 5mg twice daily vs. dalfampridine-ER 10mg twice daily: Change from baseline in EQ-5D VAS score at Visit 3; Test type: Superiority or Other; p = 0.203, ANOVA; [statistical method as in outcome 6, analysis 1]; Least Squares Mean = 2.3, 95% CI 2-sided [-1.2 to 5.8], Standard Error of Mean 1.80

ADVERSE EVENTS:
Time Frame: On or after start of double-blind treatment through 14 days after the last dose for non-serious events, or up to 30 days after the last dose for serious adverse events (SAEs).
Description: Adverse events are treatment-emergent adverse events (TEAEs) that had a date of onset or worsening, on or after start of double-blind treatment. Number of participants exposed to study medication in the Dalfampridine-ER 10mg group (142) is 1 less than total # completed. 1 patient was randomized to Dalfampridine-ER 10mg but actually received placebo
Arm/Group | Placebo | Dalfampridine-ER 5mg | Dalfampridine-ER 10mg
Serious Adverse Events (participants affected / at risk) | 0/143 | 2/144 | 2/142
Other Adverse Events (participants affected / at risk) | 77/143 | 80/144 | 84/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=143) | Dalfampridine-ER 5mg (N=144) | Dalfampridine-ER 10mg (N=142)
Breast abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Breast cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=143) | Dalfampridine-ER 5mg (N=144) | Dalfampridine-ER 10mg (N=142)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 5 (5) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5) | 6 (6)
Balance disorder (Nervous system disorders) | 6 (7) | 3 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 6 (8) | 3 (3) | 3 (3)
Dizziness (Nervous system disorders) | 3 (3) | 7 (7) | 15 (17)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 6 (7) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 7 (9) | 10 (13) | 3 (3)
Fatigue (General disorders) | 3 (3) | 4 (5) | 4 (4)
Headache (Nervous system disorders) | 16 (17) | 13 (15) | 18 (18)
Insomnia (Psychiatric disorders) | 6 (6) | 7 (7) | 11 (11)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (6) | 3 (3)
Nasopharyngitis (Infections and infestations) | 3 (3) | 2 (2) | 6 (6)
Nausea (Gastrointestinal disorders) | 5 (5) | 11 (12) | 11 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (6) | 6 (6)
Paraesthesia (Nervous system disorders) | 4 (4) | 2 (2) | 7 (12)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 5 (5) | 3 (3)
Urinary tract infection (Infections and infestations) | 8 (9) | 9 (9) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor (Acorda) has right to review and comment on proposed publications within a specified time frame, up to 60 days; multi-center trials require joint publication unless specifically permitted otherwise.